CLINICAL TRIAL: NCT06501807
Title: Real Life Assessment of Biologics Efficacy in Severe Chronic Rhinosinusitis With Nasal Polyps
Brief Title: BIOlogics in Severe Nasal POlyposis SurvEy.: a French Registry
Acronym: BIOPOSE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023_0682
Record Dates: First submitted 2024-05-21; First posted 2024-07-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Rhinosinusitis Chronic; Nasal Polyps
Keywords: nasal polyp; chronic rhinosinusitis; eosinophil; endotype
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab; mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biologic treatments available (Other): Biologic treatments available in CRSwNP (dupilumab, mepolizumab and benralizumab according to their marketing approval).
  Interventions: Drug: Biologic treatments available in Chronic Rhinosinusitis with Nasal Polyps (dupilumab, mepolizumab and benralizumab according to their marketing approval).

INTERVENTIONS:
Drug: Biologic treatments available in Chronic Rhinosinusitis with Nasal Polyps (dupilumab, mepolizumab and benralizumab according to their marketing approval). — Drug prescription according to their marketing approval (subcutaneously, every month or every two weeks).

SUMMARY:
With a prevalence of 2-4% in western countries, Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) is of major concern regarding its substantial impact on the social and physical quality of life. So far, endoscopic sinus surgery remains the treatment of choice when the first line of medical treatment with corticosteroid has failed.

During the last 15 years, several studies have shown that CRSwNP is associated with a T helper 2 (T2) immune response leading to B cell release of IgE, mucosal recruitment of eosinophils from bone marrow via Interleukin (IL)-5, IL-4 and IL-13 mediated chemoattractant production.

New biologic agents capable of blocking T2 cytokines have been developed in the field of eosinophil-associated diseases, shifting the paradigm of treatment for patients with CRSwNP. In the near future, endotype profiling with accurate biomarkers will be mandatory to tailor the treatment of nasal polyposis with specific biologic therapies.

Herein the investigators propose a prospective study monitoring medical records of CRSwNP patients who undergo biologic treatments. The objectives are to assess treatment efficacy on quality of life, to report clinical and biological criteria for prescription and to measure tolerance and compliance.Patient-reported outcomes will be addressed according to their initial clinical profile (allergy, asthma, NSAID, gastroesophageal reflux disease, obstructive apnea, otologic disorder, smoke habit).

ELIGIBILITY:
Inclusion Criteria:

* Patients of over 18-year old requiring a biologic treatment for CRswNP in accordance with its marketing approval.
* The patients already treated according to this criteria since August 2021 will be followed and their previous clinical and biological data retrospectively collected

Exclusion Criteria:

* Oral corticotherapy in the previous month;
* Biologic treatment with anti-IgE (omalizumab), anti-IL-5/IL-5R (mepolizumab, benralizumab) or anti-IL-4/IL-13R (dupilumab) or any other biotherapy for inflammatory diseases in the previous 6 months of initiation of treatment apart from ongoing biotherapies for severe asthma or CRSwNP;
* Hypersensitivity to humanized antibodies ;
* Documented SARS-Cov2 infection in the last 3 months with persistent olfactory disorders related to COVID;
* Pregnant or breast-feeding women;
* Patient without social coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2034-09-02 (Estimated); Study Completion 2035-01-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of quality of life over 5 years according to the asthmatic status of the patients | 5-year follow-up
  Assessment of disease control with the Sino-nasal outcome test-22. from 0 to 110, 110=worst outcome

SECONDARY OUTCOMES:
Quality of life progression in patients with Chronic Rhinosinusitis with Nasal Polyps | Evaluation after 6 months of treatment with biologics
  Assessment of disease control with the Sino-nasal outcome test-22. from 0 to 110, 110=worst outcome
Patient reported symptoms measurement | Month 0, Month 3, Month 6, and every 6 months until 5 years
  Number of oral corticosteroid treatment courses between each visit (in grammes)
Time to first surgical procedure since the beginning of biologic treatment | MMonth 0, Month 3, Month 6, and every 6 months until 5 years
  Date and type of sinus surgery between each visit
Blood eosinophil count and total IgE blood concentrations evolution during the course of the 5-year follow-up | Month 0, Month 3, Month 6, and every 6 months until 5 years
  Number off cells per mm3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille, Lille, France